CLINICAL TRIAL: NCT01066299
Title: A Randomized, Double-blind, Placebo-controlled Single-center Study on the Influence of Oxytocin on the Startle Reflex and on Its Modulation in Healthy Male Subjects
Brief Title: Influence of Oxytocin on the Startle Reflex and on Its Modulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: University of Basel (Other); University of Freiburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: OXT_PSY1
Record Dates: First submitted 2010-02-02; First posted 2010-02-10 (Estimated); Last update posted 2011-11-29 (Estimated); Status verified 2011-11

CONDITIONS: Psychiatric Disorders
Keywords: oxytocin; psychophysiology; startle; anxiety; emotion; physiology
MeSH Terms: conditions — Mental Disorders; Anxiety Disorders | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oxitocin nasal spray (Experimental): oxytocin nasal spray
  Interventions: Drug: Syntocinon®
- placebo (Placebo Comparator): inactive nasal spray
  Interventions: Drug: inactive nasal spray

INTERVENTIONS:
Drug: Syntocinon® — single dose of OXT (24 IU)
  Arms: oxitocin nasal spray
Drug: inactive nasal spray — single dose (24 IU)
  Arms: placebo

SUMMARY:
Oxytocin (OXT) is currently regarded as a crucial neuropeptide in the mediation of various human social behaviors, e.g. social affiliation, social recognition, and the modulation of anxiety, mood, and aggression. An impairment of social behavior, emotional regulation as well as increased stress reactions are characteristic of several psychiatric conditions, including schizophrenia, social anxiety and PTSD, in which there is also some evidence for OXT dysfunction. The startle reflex is a basic defensive reaction that can be modulated by emotional stimuli. The investigation of the startle reflex and of its modulation is a well-validated method to test stress reactions and emotional regulation. These processes are impaired in the same psychiatric diseases, in which OXT dysfunction was evidenced. Although previous animal studies showed that the dysfunction of brain OXT systems might be implicated in startle reflex and in its modulation, no study has been performed yet in human that investigated the influence of OXT administration on the startle response and on its affective modulation. A first aim of this study is to investigate the influence of OXT on stress reactivity and emotional modulation in healthy humans. A second aim is to develop a method for the investigation of anxiety disorders. Fifty male healthy participants will be tested using a randomized double-blind placebo-controlled cross-over design in two occasions; once with administration of 24 IU OXT, and once with placebo using nasal sprays while performing a computer-based experiment, in which emotional pictures and auditory startle probes are presented. We will measure the subject's subjective ratings of the pictures as well as the facial EMG activation, heart rate and electrodermal activation throughout the study. This project offers a unique opportunity to study the relationship between the OXT system and basic motivational and emotional behaviors. The investigation of these mechanisms is in turn greatly worthwhile, not only for understanding of the neurochemical and physiological processes involved in emotional regulation, but also for the comprehension of the neuroendocrine and neurophysiological mechanismsunderlying anxiety disorders. In the long term, it could open the possibilities of OXT as a psychobiological therapeutics of psychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

* gender: male
* age > 18 years
* good command of German
* non-smoker

Exclusion Criteria:

* impaired cognitive abilities
* past or current psychiatric or neurological disorder
* other relevant somatic disease (including liver, kidney or heart diseases - -- allergy to preserving agents (Paraben contained in nasal spray)
* other medication including hormonal and herbal medication
* participation in other clinical studies within one month
* impaired hearing

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Eye blink response to the tones measured as the peak activity of the left musculus orbicularis oculi that will be compared between the active drug and the placebo conditions. | 1 year

SECONDARY OUTCOMES:
Anxiety ratings assessed with the State-Trait-Inventory that will used as a covariate in the ANOVAs. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chantal Martin Soelch, PhD, Principal Investigator — University Hospital Zurich, Division of Psychiatry and Psychotherapy
Locations (1):
- University Hospital Zurich, Division of Psychiatry and Psychotherapy, Zurich, Switzerland